CLINICAL TRIAL: NCT01429909
Title: Optimization of fMRI for the Study of Basal Ganglia Activation in Parkinson's Disease: T2* Measurement in the Cortex and the Basal Ganglia
Brief Title: Optimization of fMRI for the Study of Basal Ganglia Activation in Parkinson's Disease
Acronym: 2010-A01115-34
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0097; 2010-A01115-34 (Registry Identifier: 2010-A01115-34)
Record Dates: First submitted 2011-07-07; First posted 2011-09-07 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Parkinson's Disease
Keywords: Functional magnetic resonance imaging; T2*; cortex and basal ganglia; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Device: MAGNETOM Avanto (MRI device) — The primary purpose is to optimize the fMRI by a quantitative measurement of the T2* in the cortex and the basal ganglia using MRI. The secondary purpose is to study the effect of age and Parkinson's disease on T2*.

SUMMARY:
Functional magnetic resonance imaging (fMRI) is a non-invasive imaging technique assessing neuronal activations during motor or cognitive tasks. The MRI sequences used are currently optimized for the study of cortex activations, particularly concerning the echo time (TE).Very few studies are interested in optimizing the fMRI for the study of the basal ganglia, structure implicated in many neurological diseases such as Parkinson's disease. The T2 * is a tissue parameter dependent of iron content, which differs with brain structures and probably also with age and in case of neurodegenerative disease. Optimal TE s should correspond to the T2 * of studied brain structure The primary purpose is to optimize the fMRI by a quantitative measurement of the T2* in the cortex and the basal ganglia using MRI. The secondary purpose is to study the effect of age and Parkinson's disease on T2*.

DETAILED DESCRIPTION:
80 subjects (40 PD patients and 40 paired healthy volunteers (on sex and age)) aged 40-80 years will be included. PD patients will be recruited in the Department of Neurology of CHU of Clermont-Ferrand. Healthy volunteers will be selected in clinical trial database. This study will consist of one visit (at J0) during which subjects will undergo a MRI (a single acquisition of 40 minutes approximately). PD patients will be further questioned on their disease and will benefit from a neurological examination

ELIGIBILITY:
Inclusion Criteria:

* For patients :
* Patients with idiopathic Parkinson's disease according to UKPDSBB criterias
* Men or women aged between 40 to 80 years
* not treated with deep brain stimulation

For healthy subjects

- Men or women aged between 40 to 80 years

Exclusion Criteria:

For patients

* Dementia (MMS<24)
* Contraindication to MRI.
* Under guardianship
* In excluding period for another study

For healthy subjects

* Antecedent of neurodegenerative diseases or psychiatric diseases
* Contraindication to MRI
* Under guardianship
* In excluding period for another study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The quantitative measurement of T2* in the cortex and basal ganglia using MRI, made à J0. | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Miguel ULLA, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France